CLINICAL TRIAL: NCT04379297
Title: COvid-19 National Survey for Assessing VIral Spread by Nonaffected CarriErs (CON-VINCE)
Acronym: CON-VINCE
Status: Completed | Type: Observational
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Luxembourg National Research Funds (Unknown); University of Luxembourg (Other); Centre Hospitalier du Luxembourg (Other); TNS-Ilres (Unknown); Laboratoires Réunis (Unknown); BioneXt Lab (Unknown); Ketterthill (Unknown); Laboratoire National de santé (Unknown)
Responsible Party: Sponsor
Other Study IDs: CNER 202004/01; 831x6ce0d (Other: Ministry of Health); FNR/CON-VINCE (Other Grant/Funding Number: Luxembourg National Research Fund)
Record Dates: First submitted 2020-05-06; First posted 2020-05-07 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: COVID19
Keywords: Coronavirus; COVID; Prevalence
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Naso-pharyngeal swab, Oro-pharyngeal swab, Blood, sputum,Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CON-VINCE (COvid-19 National survey for assessing VIral spread by Non-affected CarriErs) is a national, monocentric, and longitudinal study aiming to evaluate the spread dynamics of the COVID-19 disease within the Luxembourgish population. Participants who are clinically asymptomatic or present with only mild symptoms will be followed up longitudinally, regularly tested for SARS-CoV-2 by RT-PCR, antibody status, and subjected to an epidemiological, clinical and biological phenotyping to better understand the nature, dynamics of infectivity and spread of the virus in the population. CON-VINCE will also track the psychological and socio-economic impact of long-term containment measures on the general population.

DETAILED DESCRIPTION:
To capture the dynamics and impact of the virus spread in the Luxembourgish population, data and sample collection is done every two weeks for two months (4 times in total) with a final follow-up one year after the participant's inclusion in the study. Participants complete questionnaires before each sample collection. The baseline questionnaire captures demographic data, medical history, behavioral and psychological data, and socio-economic status. Participants provided information on medical history, history of allergies, smoking, and chronic medication taken regularly. COVID-19-related data and environmental conditions of the household were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 and older of both genders, with a full capacity of consent.
* SARS-CoV-2-positive individuals with an asymptomatic or oligosymptomatic infection (mild or oligosymptomatic disease course is defined as absence of fever and respiratory distress or cough not attributable to other known chronic disease).
* OR SARS-CoV-2-negative individuals at the time of inclusion.
* OR post-infectious SARS-CoV-2-negative individuals with acquired immunity to SARS-CoV-2 and a mild disease course.

Exclusion Criteria:

* Evolution of the COVID-19 disease requiring a hospital admission before inclusion in the study
* Presence of fever and respiratory distress/cough at the time of inclusion not attributable to other known chronic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Representative panel of the Luxembourgish population
Sampling Method: Probability Sample
Enrollment: 1870 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence and dynamics of the SARS-COV 2 infection in Luxemburg | 04.2020-05.2021
  Evaluation of the prevalence by RT-PCR and serology testing
Collection of samples for research | 04.2020-05.2021
  Samples will be analysed and stored for future research

SECONDARY OUTCOMES:
Psycho-social evaluation | 04.2020-05.2021
  Psychological and socio- economic impact of long-term containment measures on the general population

CONTACTS AND LOCATIONS:
Overall Officials: Rejko Krüger, Dr, Principal Investigator — Luxembourg Institute of Health
Locations (1):
- Luxembourg Institute of Health, Strassen, Luxembourg

REFERENCES:
- [Result] Tsurkalenko O, Bulaev D, O'Sullivan MP, Snoeck C, Ghosh S, Kolodkin A, Rommes B, Gawron P, Rauschenberger A, Moreno CV, Gomes CPC, Kaysen A, Ohnmacht J, Schroder VE, Pavelka L, Meyers GR, Pauly L, Pauly C, Hanff AM, Meyrath M, Leist A, Sandt E, Aguayo GA, Perquin M, Gantenbein M, Abdelrahman T, Klucken J, Satagopam V, Hilger C, Turner J, Vaillant M, Fritz JV, Ollert M, Kruger R; CON-VINCE consortium and the ORCHESTRA working group. Creation of a pandemic memory by tracing COVID-19 infections and immunity in Luxembourg (CON-VINCE). BMC Infect Dis. 2024 Feb 9;24(1):179. doi: 10.1186/s12879-024-09055-z. PMID 38336649
- [Result] Ribeiro F, Schroder VE, Kruger R, Leist AK; CON-VINCE Consortium. The evolution and social determinants of mental health during the first wave of the COVID-19 outbreak in Luxembourg. Psychiatry Res. 2021 Sep;303:114090. doi: 10.1016/j.psychres.2021.114090. Epub 2021 Jun 30. PMID 34247057